CLINICAL TRIAL: NCT05808673
Title: A Randomized, Double-blind, Parallel Controlled, Phase I Three-arm Study, Comparing the PK, PD, Safety, and Immunogenicity of Pre- and Post-change CMAB807X, Post-change CMAB807X and Xgeva® in Healthy Chinese Male Subjects
Brief Title: Study of CMAB807X Pre- and Post-change in Manufacturing Site and Xgeva® in Healthy Volunteers
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Changes in the company's production plan
Sponsor: Taizhou Mabtech Pharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMAB807X-001
Record Dates: First submitted 2023-03-27; First posted 2023-04-11 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2023-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Denosumab

STUDY DESIGN:
Intervention Model Description: Biological: Pre- and Post-change CMAB807X, Xgeva®
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Post-change CMAB807X (Experimental): 120 mg Subcutaneous injection around belly button
  Interventions: Biological: Post-change CMAB807X
- Pre-change CMAB807X (Other): 120 mg Subcutaneous injection around belly button
  Interventions: Biological: Pre-change CMAB807X
- Xgeva® (Active Comparator): 120 mg Subcutaneous injection around belly button
  Interventions: Biological: Xgeva®

INTERVENTIONS:
Biological: Post-change CMAB807X — for subcutaneous injection only
  Arms: Post-change CMAB807X
Biological: Pre-change CMAB807X — for subcutaneous injection only
  Arms: Pre-change CMAB807X
Biological: Xgeva® — for subcutaneous injection only
  Arms: Xgeva®

SUMMARY:
This is a randomized, double-blinded, controlled Phase I three-arms study of CMAB807X administered by subcutaneous injection. This study will characterize the pharmacokinetic, pharmacodynamics, safety and immunogenicity of CMAB807X Pre- and Post-change in Manufacturing Site, and Post-change CMAB807X versus Xgeva® #Denosumab# in healthy male subjects after a single dose

DETAILED DESCRIPTION:
This is a randomized, double-blind, parallel-controlled, single-dose phase I three-arms clinical study in healthy Chinese male subjects. A total of 252 subjects were planned to be enrolled and randomly assigned to the test group or the bridging control group or bioequivalence control group in a 1:1:1 ratio. Subjects in three groups received a single abdominal subcutaneous injection of pre- or post-change CMAB807X or Xgeva® #Denosumab# 120 mg, respectively. Subjects in three groups were observed for 140 days after administration to evaluate similarities in pharmacokinetics, pharmacodynamics, safety, and immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteers, age ranged 18 to 45 years (both inclusive) when sign the informed consent form.
2. Subjects with body weight of ≥58 kg and ≤ 68 kg and BMI ≥18 and ≤ 28 kg/m2.
3. Subjects were willing to take effective contraceptive measures throughout the study period (including: physical contraception, surgery, abstinence, etc.,) until at least 6 months after administration.
4. Subjects have the ability to understand the full characteristics and objectives of the study, including the possible risks and side effects of the study; moreover, subjects can communicate well with researchers and complete the research according to the regulations.
5. Subjects must be informed consent of the study and voluntarily sign ICF (name and time) prior to the study.

Exclusion Criteria:

1. After medical examination (vital signs, physical examination, electrocardiogram, chest X-radiography, cervical and abdominal B-ultrasound, and various laboratory examinations including blood routine, urine routine, blood biochemistry, etc.), any examination item was judged abnormal by the investigator and had clinical significance.
2. Serum calcium level were out of the normal range.
3. QTcF > 450 ms (12-lead ECG).
4. Inflammation or abnormalities in or around the site of administration.
5. Those who have a history of serious diseases including but not limited to nervous system, cardiovascular system, blood and lymphatic system, immune system, urinary system, digestive system, respiratory system, metabolic and skeletal systems, or currently have any of the above diseases or active infected diseases, or any other disease or medical condition that may interfere with the results of the trial, such as hereditary bleeding tendency, coagulation disorders or history of blood clots or bleeding.
6. Previous diagnosis of bone disorders that the investigator has determined to be clinically significant, or any disease that affects bone metabolism, including but not limited to: malignant tumors (including myeloma), hypothyroidism/hyperthyroidism, hypoparathyroidism/hyperthyroidism, acromegaly, Cushing's syndrome, hypopituitarism, severe chronic obstructive pulmonary disease, rheumatoid arthritis, osteomalacia, etc.
7. Subjects with past or current osteomyelitis or osteonecrosis of the jaw (ONJ), or risk factors for ONJ, such as dental disease or jaw disease requiring oral surgery, dental surgery; or plan to have dental surgery during the study.
8. Fracture occurred within 6 months prior to signing ICF.
9. Surgery within 6 months prior to signing ICF, or plan to have surgery during the study period.
10. Allergic to two or more drugs or foods, or to any component of the investigational agent.
11. Use of any prescription drug, over-the-counter drug, vitamin or herbal medicine within 30 days prior to signing ICF, or prior use of drugs within 5 half-lives, whichever is longer.
12. Use of any medications that have the potential to affect bone metabolism prior to administration (e.g., bisphosphonate or fluoride, estrogen, selective estrogen receptor modulators, calcitonin, parathyroid hormone, high-dose vitamin D (> 1000 IU/ day), anabolic steroids, systemic glucocorticoids, or percalcitriol within 6 months)
13. Use of anti-RANKL mab within 12 months, or any biological agent within 3 months prior to signing ICF.
14. Those who have received vaccine within the 4 weeks prior to signing ICF, or who plan to receive live vaccine during the study period.
15. History of drug abuse, or positive urine drug screening.
16. Those who had donated or lost blood at least 200 mL in the 3 months prior to signing ICF, or planned to donate blood during the study.
17. Those who can not tolerate venipunction, has a history of dizziness of needle and blood.
18. Those who have been enrolled in other drug or device clinical studies within 3 months prior to signing ICF.
19. Those who smoked more than 5 cigarettes per day in the 6 months prior to signing ICF and did not cooperate with smoking bans during the study period.
20. Those who consumed more than 14 units of alcohol per week (1 unit = 17.7mL ethanol, i.e., 1 unit = 357mL 5% beer or 43mL 40% liquor or 147mL 12% wine) in the 3 months prior to signing ICF, or not willing to ban alcohol during the study period.
21. Those who excessively daily consumed tea, coffee or caffeinated beverages (more than 8 cups, 1 cup =250mL) in the 3 months prior to signing ICF.
22. Those who have special dietary requirements, or can not accept uniform diet
23. Other conditions considered inappropriate to be included in this study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-time Curve From Zero (0) Hours Extrapolated to infinite time | up to 3336 hours
  Area Under the Plasma Concentration-time Curve From Zero (0) Hours Extrapolated to infinite time After the Single injection of Denosumab
Maximum Concentration of Denosumab | up to 3336 hours
  Maximum Concentration of Denosumab After the Single Injection of denosumab

SECONDARY OUTCOMES:
Time to Maximum Concentration of Denosumab | up to 3336 hours
  Time to Maximum Concentration of Denosumab after the Single Injection of
Area Under the Plasma Concentration-time Curve From Zero (0) Hours to 3336 Hours | up to 3336 hours
  Area Under the Plasma Concentration-time Curve From Zero (0) Hours to 3336 Hours After the Single Injection of Denosumab
Half time | up to 3336 hours
  Half-time after the Single Injection of Denosumab
Clearance Rate | up to 3336 hours
  Clearance Rate after the Single Injection of Denosumab
Apparent Volume of Distribution | up to 3336 hours
  Apparent Volume of Distribution after the Single Injection of Denosumab
Serum type 1 C-telopeptide (CTX1) | up to 3336 hours
  CTX1 level in the serum samples from subjects
anti-drug antibodies(ADA) | up to 3336 hours
  ADA Positive Rate after the Single Injection of Denosumab
Neutralization antibodies(Nab) | up to 3336 hours
  Neutralizing Antibody Positive Rate after the Single Injection of Denosumab

OTHER OUTCOMES:
Percentage and Severity of Participants with Adverse Events | up to 3336 hours
  Total Frequency and Severity of Adverse Events/Serious Adverse Events Within the Whole Time of the Study

CONTACTS AND LOCATIONS:
Overall Officials: Hu Wei, Doctor, Principal Investigator — The Second Hospital of Anhui University
Locations (1):
- The Second Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No